CLINICAL TRIAL: NCT02290912
Title: Gray Matters: Multi-domain Lifestyle Behavioral Alzheimer's Disease Prevention Randomized Controlled Trial
Brief Title: Gray Matters Alzheimer's Disease Prevention Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Maria C Norton, PhD, Professor, Utah State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5606
Record Dates: First submitted 2014-11-06; First posted 2014-11-14 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease prevention lifestyle intervention
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Health education program; informational website, experiential classes in various help domains, custom smart phone application, and wearable technology
  Interventions: Behavioral: Health education program
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Health education program — The intervention is a health education program including: informational website, experiential classes, custom smart phone or smart table application, wearable activity monitor, and informal coaching by student researchers to provide moral support for lifestyle behavioral change goals. Participants are not placed on any specific behavioral regimen but instead are encouraged to adopt healthier lifestyle behaviors per the evidence-based health education program, and to attend the experiential classes "cafeteria style" (i.e. based on their individual preferences).
  Arms: Treatment

SUMMARY:
This is a randomized controlled trial to develop and test the efficacy of a multi-domain lifestyle behavioral intervention designed to promote healthier lifestyle behaviors linked to lower Alzheimer's disease risk among persons aged 40 to 64 years.

DETAILED DESCRIPTION:
This is a randomized controlled trial to develop and test the efficacy of a multi-domain lifestyle behavioral intervention designed to promote healthier lifestyle behaviors linked to lower Alzheimer's disease risk among persons aged 40 to 64 years. Participants are randomized to treatment or control condition. The intervention, spanning a six month period, is an evidence-based health education program.

ELIGIBILITY:
Inclusion Criteria:

* Age
* Residing or working in Cache County Utah
* Possessing smart phone or tablet

Exclusion Criteria:

* Dementia
* Pregnancy
* Untreated chronic major depression or other psychiatric condition
* Body mass index > 41
* Heart or stroke in prior 6 weeks
* Active cancer treatment
* Unwillingness to seek medical help when serious condition identified at intake

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Picture Vocabulary | up to 7 months
  Picture Vocabulary cognitive test score
Flanker Inhibitory Control and Attention Test | up to 7 months
  Flanker Inhibitory Control and Attention Test cognitive test score
List Sorting Working Memory Test | up to 7 months
  List Sorting Working Memory Test cognitive test score
Oral Symbol Digit Test | up to 7 months
  Oral Symbol Digit Test cognitive test score
Montreal Cognitive Assessment | up to 7 months
  Montreal Cognitive Assessment test score
Rey Auditory Verbal Learning Test | up to 7 months
  Rey Auditory Verbal Learning Test score
Controlled Oral Word Association Test | up to 7 months
  Controlled Oral Word Association Test score
Blood pressure | up to 7 months
  Systolic and diastolic blood pressure
Body mass index | up to 7 months
  Height and weight measurement for computing body mass index
Insulin | up to 7 months
  insulin from venipuncture blood sample
Systemic inflammation | up to 7 months
  C-reactive protein from venipuncture blood sample
Skin carotenoid status | up to 7 months
  Biophotonic device that shines a light-emitting diode (LED) light at a site on the palm, to measure the skin carotenoid level in units of Raman counts
Triglycerides | up to 7 months
  triglycerides from venipuncture blood sample
HDL Cholesterol | up to 7 months
  High-density lipoprotein from venipuncture blood sample
LDL Cholesterol | up to 7 months
  Low-density lipoprotein from venipuncture blood sample
Total cholesterol | up to 7 months
  Total cholesterol from venipuncture blood sample

SECONDARY OUTCOMES:
Depression | up to 7 months
  Center for Epidemiologic Studies - Depression scale score
Motivation | up to 7 months
  Situational Motivation Scale score
Sleep Quality | up to 7 months
  Pittsburgh Sleep Quality Index scale score
Stress | up to 7 months
  Perceived Stress Scale score
Emotional Support | up to 7 months
  Emotional Support subscale from the NIH Toolbox measures for social engagement
Friendship | up to 7 months
  Friendship subscale from the NIH Toolbox measures for social engagement
Hostility | up to 7 months
  Hostility subscale from the NIH Toolbox measures for social engagement
Loneliness | up to 7 months
  Loneliness subscale from the NIH Toolbox measures for social engagement
Physical Activity - Moderate | up to 7 months
  self-report question concerning # minutes per day doing moderate intensity physical activity (per Center for Disease Control definition)
Physical Activity - Vigorous | up to 7 months
  self-report question concerning # minutes per day doing vigorous intensity physical activity (per Center for Disease Control definition)
Nutrition | up to 7 months
  Diet History Questionnaire
Readiness for Change | up to 7 months
  Revised University of Rhode Island Change Assessment (R-URICA) readiness for change scale
Metacognition | up to 7 months
  Total score from a set of seven items (1=much worse to 5=much better), comparing current memory to how it was three years ago, adapted from a questionnaire of functional ability

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Norton, PhD, Principal Investigator — Utah State University

REFERENCES:
- [Derived] Hartin PJ, Nugent CD, McClean SI, Cleland I, Tschanz JT, Clark CJ, Norton MC. The Empowering Role of Mobile Apps in Behavior Change Interventions: The Gray Matters Randomized Controlled Trial. JMIR Mhealth Uhealth. 2016 Aug 2;4(3):e93. doi: 10.2196/mhealth.4878. PMID 27485822